CLINICAL TRIAL: NCT07112755
Title: Development of a Risk Prediction Model for Osteopenia in Patients With Psoriasis: A Cross-Sectional Study
Brief Title: Prediction Model for Osteopenia in Patients With Psoriasis
Status: Completed | Type: Observational
Sponsor: Chongli Yu (Other)
Responsible Party: Sponsor-Investigator, Chongli Yu, PhD Candidate, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: S2022-196-01-01
Record Dates: First submitted 2025-08-02; First posted 2025-08-08 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Psoriasis
Keywords: psoriasis; osteopenia
MeSH Terms: conditions — Psoriasis; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to develop a clinical prediction model for osteopenia in patients with psoriasis. By retrospectively analyzing demographic, laboratory, and lifestyle variables, the investigators will identify risk factors associated with decreased bone mineral density (BMD) in this population. The study will facilitate the identification of high-risk individuals and provide evidence for early screening and intervention strategies.

DETAILED DESCRIPTION:
Psoriasis is a chronic inflammatory skin disease associated with various systemic comorbidities, including an increased risk of bone loss. Recent studies suggest that patients with psoriasis have a significantly higher incidence of osteopenia and osteoporosis than the general population, potentially due to systemic inflammation and shared risk factors. All enrolled patients will undergo dual-energy X-ray absorptiometry (DEXA) scans to assess bone mineral density (BMD). Based on the results, patients will be categorized into normal BMD and osteopenia groups. Demographic data (age, sex, height, weight, BMI), clinical variables (disease duration, CRP, ESR, blood glucose, blood lipids, blood pressure), and lifestyle factors (smoking, alcohol use) will be collected and analyzed. Univariate and multivariate logistic regression analyses will be performed to identify independent risk factors. A prediction model will be constructed and evaluated using ROC curve analysis to assess sensitivity, specificity, and accuracy. The objective of this study is to develop a validated tool to assist clinicians in identifying patients with psoriasis at high risk for osteopenia, thereby enabling early screening and preventive management to reduce future fracture risk.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of plaque psoriasis according to established diagnostic criteria
* Age ≥ 18 years
* Willingness to participate in the study and provide written informed consent

Exclusion Criteria:

* Severe hepatic or renal dysfunction
* Coexisting immune, endocrine, or malignant diseases that may affect bone metabolism
* Congenital joint deformities, history of joint trauma, or joint replacement surgery
* Use of systemic corticosteroids, calcium supplements, or bisphosphonates within the past 3 months
* Psychiatric or psychological disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with plaque psoriasis who attended the Department of Dermatology at the First Medical Center of the PLA General Hospital. Eligible participants were aged 18 years or older and underwent bone mineral density assessment by DEXA. Patients with significant comorbidities affecting bone metabolism were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Occurrence of Osteopenia in Patients With Psoriasis | At the time of DEXA assessment during enrollment
  Bone mineral density (BMD) will be assessed using dual-energy X-ray absorptiometry (DEXA) at the lumbar spine and/or femoral neck. Osteopenia is defined as a T-score between -1.0 and -2.5 according to WHO criteria. Patients will be categorized accordingly.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hosptial, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sirufo MM, De Pietro F, Bassino EM, Ginaldi L, De Martinis M. Osteoporosis in Skin Diseases. Int J Mol Sci. 2020 Jul 3;21(13):4749. doi: 10.3390/ijms21134749. PMID 32635380
- [Background] Ogdie A, Harter L, Shin D, Baker J, Takeshita J, Choi HK, Love TJ, Gelfand JM. The risk of fracture among patients with psoriatic arthritis and psoriasis: a population-based study. Ann Rheum Dis. 2017 May;76(5):882-885. doi: 10.1136/annrheumdis-2016-210441. Epub 2017 Jan 16. PMID 28093419
- [Background] Sepehri NZ, Raeisi T, Razi B, Janmohammadi P, Darand M, Alizadeh S. The association between psoriasis and psoriatic arthritis with the risk of osteoporosis, osteopenia and bone fractures: A systematic review and meta-analysis. Int J Clin Pract. 2021 Nov;75(11):e14630. doi: 10.1111/ijcp.14630. Epub 2021 Jul 22. PMID 34260133
- [Background] D'Epiro S, Marocco C, Salvi M, Mattozzi C, Luci C, Macaluso L, Giancristoforo S, Campoli M, Scarno M, Migliaccio S, Calvieri S, Richetta A. Psoriasis and bone mineral density: implications for long-term patients. J Dermatol. 2014 Sep;41(9):783-7. doi: 10.1111/1346-8138.12546. Epub 2014 Jul 3. PMID 24990650
- [Background] Ojeda JL, Ros MA, Garcia-Porrero JA. [Role of the basement membrane in the pathogenesis of polycystic kidney: a new pathogenetic hypothesis based on an experimental model]. Minerva Urol Nefrol. 1987 Jul-Sep;39(3):275-82. No abstract available. Italian. PMID 3326187
- [Background] Ding X, Wang T, Shen Y, Wang X, Zhou C, Tian S, Liu Y, Peng G, Zhou J, Xue S, Wang R, Tang Y, Meng X, Pei G, Bai Y, Liu Q, Li H, Zhang J. Prevalence of psoriasis in China: a population-based study in six cities. Eur J Dermatol. 2012 Sep-Oct;22(5):663-7. doi: 10.1684/ejd.2012.1802. PMID 22910173